CLINICAL TRIAL: NCT06975150
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Group, 12 Weeks, Phase 2b Clinical Study to Evaluate the Efficacy and Safety of HK-660S in Patients With Primary Sclerosing Cholangitis (PSC)
Brief Title: Efficacy and Safety of HK-660S in the Treatment of Primary Sclerosing Cholangitis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: CuromeBiosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HK-660S-202
Record Dates: First submitted 2025-05-08; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Primary Sclerosing Cholangitis (PSC)
Keywords: HK-660S-202; PSC; Primary Sclerosing Cholangitis; HK-660S
MeSH Terms: conditions — Cholangitis, Sclerosing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind (Participant, Investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- HK-660S 100mg (Experimental): oral administration of 100 mg HK-660S (one active tablet and one placebo tablet) twice a day on an empty stomach in the morning and evening
  Interventions: Drug: HK-660S 100mg
- HK-660S 200mg (Experimental): oral administration of 200 mg HK-660S (two active tablets) twice a day on an empty stomach in the morning and evening
  Interventions: Drug: HK-660S 200mg
- Placebo (Placebo Comparator): oral administration of two placebo tablets twice a day on an empty stomach in the morning and evening
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HK-660S 100mg — Administered orally
  Arms: HK-660S 100mg
Drug: HK-660S 200mg — Administered orally
  Arms: HK-660S 200mg
Drug: Placebo — Administered orally
  Arms: Placebo

SUMMARY:
The cause of PSC is unknown.To date, there is no treatment besides liver transplantation proven to improve PSC prognosis. However, there is a clear medical unmet need yet for patients with PSC, due to risks and complications of liver transplantation.

This is a two-part, Phase 2b, randomized, double-blind, placebo-controlled study designed to assess the efficacy and safety of HK-660S in patients with PSC.

The primary objective is to evaluate the effects of HK-660S on serum ALP improvement (reduction of 20% or more) over 12 weeks of treatment in patients with PSC.

DETAILED DESCRIPTION:
This is a two-part, Phase 2b, randomized, double-blind, placebo-controlled study designed to assess the efficacy and safety of HK-660S in patients with PSC.

After subjects voluntarily consent in writing to participate in the clinical study, subjects who meet the inclusion/exclusion criteria will be evaluated through a screening period. The screening period should not, as far as possible, exceed a maximum of 5 weeks including the washout period. Based on the screening results at Visit 1, subjects suitable for participation in this clinical study will be selected.

In Part A, 6 subjects will be assigned to 200 mg HK-660S twice a day for 12 weeks. After Visit 2, subjects will visit the study center at Week 4 (Visit 3), Week 8 (Visit 4), Week 12 (Visit 5 / End of Treatment), and Week 16 (Visit 6 / Follow-up) to assess the efficacy and safety (excluding MRCP at Visit 6). Enrollment will be staggered, with the first two subjects enrolled and monitored for the initial 4-week treatment period. Interim safety data from these initial two subjects will be reviewed by the Sponsor and medical monitor to assess any significant safety concerns. If no such concerns are identified, enrollment of the remaining four subjects will proceed. Safety data from the first 4-week treatment in all 6 subjects will be reviewed by the SRC, which will decide on the initiation of Part B.

In Part B, 99 subjects will be randomly assigned in a 1:1:1 ratio into one of three groups: 100 mg HK-660S, 200 mg HK-660S, or placebo to take two tablets (1 active and 1 placebo tablets, 2 active tablets, or 2 placebo tablets) twice a day for 12 weeks. After Visit 2, subjects will visit the study center at Week 4 (Visit 3), Week 8 (Visit 4), Week 12 (Visit 5 / End of Treatment), and Week 16 (Visit 6 / Follow-up) to assess the efficacy and safety (excluding MRCP at Visit 6).

The study period for each subject is approximately 21 weeks including up to 5-week screening period, 12-week treatment period, and 4-week follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged ≥ 18 years.

   * Subjects and their sexual partner(s) who do not plan to become pregnant and agree to use at least one effective, appropriate contraceptive method (defined below) during the study period and up to 30 days after the last dosing of study drug
   * Contraception method: 1) hormonal contraceptives, 2) intrauterine contraceptive device or implantation of intrauterine system, 3) double-barrier method (combined use of spermicides and condoms, diaphragm, contraceptive sponge, or FemCap), or 4) sterilization (e.g., vasectomy, tubal ligation)
   * Women who are post-menopausal (have amenorrhea for 12 months or over 6 weeks after bilateral oophorectomy) and unlikely to become pregnant
2. Subjects who have a diagnosis of PSC:

   * Serum alkaline phosphatase (ALP) of > 2.0 x upper limit of normal (ULN) at screening
   * Subjects who have sclerosing cholangitis due to multifocal bile duct in magnetic resonance cholangiopancreatography (MRCP) or endoscopic retrograde cholangiopancreatography (ERCP) within 6 months from screening
3. Subjects who are able to understand information provided directly or via his/her representative and to give voluntary, written consent to participate in the study.

Exclusion Criteria:

1. Subjects with an average alcohol intake of more than 20g per day within 2 years prior to screening.
2. Subjects who have a diagnosis of type 1 diabetes or uncontrolled type 2 diabetes (HbA1c ≥ 9%) prior to screening.
3. Subjects who have chronic liver diseases other than PSC: non-alcoholic fatty liver disease, viral chronic hepatitis, alcoholic liver disease, primary biliary liver cholangitis, biliary obstruction, autoimmune hepatitis, hemoglobin deposition, Wilson's disease, α-1 antitrypsin deficiency, etc.
4. Subjects who have a diagnosis of primary biliary cholangitis or secondary sclerosing cholangitis in MRCP or ERCP prior to screening.
5. Subjects who have obstacles to MRCP implementation (e.g., cardiac pacemakers, clipped cerebral aneurysms, metallic foreign objects in the eyeball, claustrophobia).
6. Subjects who have ALT or AST > 5 x ULN.
7. Subjects who have serum creatinine ≥ 2 mg/dl.
8. Subjects who are deemed unsuitable for participation in the study at Screening, at the discretion of the investigator, due to the following: cirrhosis, severe metabolic disease, severe renal failure, severe lung disease, severe neuro/psychiatric disease, muscle disease, etc.
9. Subjects who have any clinically significant cardiovascular diseases.
10. Subjects who have uncontrolled thyroid diseases including hyperthyroidism and hypothyroidism. However, subjects who have been stably managed with thyroid disease treatment for at least 6 months prior to Screening may be included at the discretion of the investigator.
11. Subjects who have a history of immune diseases: autoimmune thrombocytopenic purpura, systemic lupus erythematosus, autoimmune hemolytic anemia, severe psoriasis, rheumatoid arthritis, etc. However, at the discretion of the investigator, patients with atopic dermatitis that is mild or can be stably managed with topical atopic dermatitis treatment may be included.
12. Subjects who had bariatric surgery within 6 months prior to screening.
13. Subjects who have undergone or are planned for liver transplantation or with current model of end stage liver disease (MELD).
14. Subjects who have positive results at the Screening visit for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV).
15. Subjects who have a history of chronic infections or have severe or life-threatening infections, or symptoms that may be considered related to infections (e.g., fever, cough). However, subjects with mild-to-moderate inflammatory bowel diseases (e.g., ulcerative colitis, Crohn's disease) who can be stably managed with 5-aminosalicylic acid, azathioprine or topical steroids may be included at the discretion of the investigator. Subjects on biologics (e.g. infliximab, adalimumab, vedolizumab, ustekinumab) or JAK inhibitors (e.g. tofacitinib) for IBD treatment are allowed if the dose has been stable for at least 12 weeks before Screening and is expected to remain stable throughout the study.
16. Subjects with evidence of an active infection during the screening period.
17. Subjects diagnosed with a malignant tumor without complete cure within 5 years prior to screening.
18. Subjects whose medication history includes any of the following drugs, within a period of 5 times the half-life of the respective drug prior to screening:

    * Therapeutics agents for steatohepatitis: thiazolidinediones, high-dose vitamin E (800 IU/day), pentoxifylline
    * Medications possibly related to PSC: high-dose ursodeoxycholic acid (UDCA; doses smaller than 28 mg/kg/day may be permitted if administered stably without change in dosage from 3 months prior to screening), immunosuppressants, obeticholic acid (OCA), budesonide, docosahexaenoic acid, methotrexate, metronidazole, minocycline, mycophenolate mofetil, nicotine, pentoxifylline, pirfenidone, prednisolone, systemic glucocorticoids, tacrolimus (If a patient is on any of the following medications and/or supplements, he or she can participate only expected to remain on the same daily dose through the treatment period: UDCA, vancomycin, azathioprine, prednisone [or an equivalent steroid compound]).
19. Subjects who administered herbal medicine or folk remedies to improve fatty liver disease within 2 weeks prior screening.
20. Subjects who have a history of alcohol or drug abuse within 5 years prior to screening.
21. Subjects who have a hypersensitivity to any excipients of the study drug.
22. Subjects who participated in another drug trial within 30 days prior to screening.
23. Subjects who are considered inappropriate to participate in clinical trials at the discretion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2025-08-18 (Estimated); Primary Completion 2028-08-30 (Estimated); Study Completion 2028-08-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects who show improvement of ALP | 12 weeks from baseline
  The improvement of ALP is defined as 20% or more ALP reduction

SECONDARY OUTCOMES:
Percentage of subjects who show improvement of severity of PSC | 12 weeks from baseline
  The improvement of severity is defined as a decrease of -1 or more in the MRCP Anali score
Percentage of subjects who show improvement of bile duct strictures in MRCP | 12 weeks from baseline
  Defined as improvement (absence or improvement) in at least one of bile strictures, dilatation or bile ductal wall thickening and enhancement based on the IPSCSG (International Primary Sclerosing Cholangitis Study Group) MRI Reporting Guideline.
Percentage of subjects who show 50% or more reduction of ALP | 12 weeks from baseline
Percentage of subjects who show ALP normalization or partial normalization (< 1.5 x ULN) | 12 weeks from baseline
Percentage of subjects who show improvement of severity of fibrosis in FibroScan | 12 weeks from baseline
Change of fibrosis score in FibroScan | 12 weeks from baseline
Percentage of subjects who show improvement of severity of liver fibrosis in Enhanced Liver Fibrosis (ELF) score | 12 weeks from baseline
Change of ELF score | 12 weeks from baseline
Change of pruritus score | 4, 8, and 12 weeks from baseline
Change of serum C4 (7α-hydroxy-4-cholesten-3-one) level | 12 weeks from baseline
Change of ALP level | 4, 8, and 12 weeks from baseline
Change of ALT, AST, GGT, and bilirubin levels | 4, 8, and 12 weeks from baseline

IPD SHARING:
Plan to Share IPD: Undecided